CLINICAL TRIAL: NCT05802758
Title: Compassion-focused Mental Health Intervention With Exposure Training in Virtual Reality for Youngsters Living in an Institution
Brief Title: CFT-focused Mental Health Intervention With Exposure Training for Youngsters
Acronym: CFT+VR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Nina Lindberg, senior doctor, professor, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS/345/2023
Record Dates: First submitted 2023-03-25; First posted 2023-04-07 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Conduct Disorder; Psychopathic Personality Trait
Keywords: psychotherapy, virtual reality, boys
MeSH Terms: conditions — Conduct Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Youngsters who get CFT + VR (Active Comparator): yougsters, who get compassion-focused short intervention together with training in virtual reality together with general psychosocial rehabilitation offered by prisons and state residential schools
  Interventions: Behavioral: Psychopathy.comp and training in virtual reality (VR)
- Treatment as usual (No Intervention): youngsters, who get only general psychosocial rehabilitation offered by prisons and state residential schools

INTERVENTIONS:
Behavioral: Psychopathy.comp and training in virtual reality (VR) — Psychopathy.comp is a CFT-based manualized program of 20 sessions a 60 min, on a weekly basis. During the CFT-intervention, partipants try out their new skills in a tailored VR setting (x5)
  Arms: Youngsters who get CFT + VR

SUMMARY:
The aim of this study is to explore if individual CFT-based intervention with exposure training in virtual reality decreases conduct disorder symptoms and callous-unemoitonal traits , as well as increases subjective emotional welbeing among 15-to-20 year-old male prisoners and boys placed to state's residential schools. We will also study factors that may predict adherence to the intervention. These factors include mental well-being, motivation, and working alliance. In addition, we will evaluate the costs of the program.

ELIGIBILITY:
Inclusion Criteria:

* Express conduct disorder psychopathology and psychopathic personality traits
* Are placed to a prison or a state residential school for at least 9 months

Exclusion Criteria:

* Females
* Non-Finninsh-speaking
* Remaining in the institution facility less than 9 months
* Intellectual dissability
* Presence of psychotic symptoms
* Autism
* History of epilepsy
* Currently participating another psychotherapeutic intervention

Ages: 15 Years to 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The self-reported change in Youth Pysychopathic traits Inventory- short version (YPI-S) and in the factors of it | 5 months
  Measures both conduct prolems and psychopathic traits

SECONDARY OUTCOMES:
Short Warwick-Edinburgh Wellbeing scale (SWEMWBS) | 5months
  measures general psychosocial well-being
Difficulties in Emotion Regulating Scale-Short form (DERS-SF) | 5 months
  measures emotion regulation style
WHO's quality of life questionnaire- Brief version (WHOQOL-BREF) | 5 months
  measures quality of life
Self-Compassion Scale- Short Form (SCS-SF) | 5 months
  measures self-compassion
Santa Clara Compassion Scale | 5 months
  masures compassion against other people
Young Person's Clinical Outcomes in Routine Evaluation (YP-CORE) | 5 months
  measures how the intervention is felt by the youngster
Situational intrinsic and extrinsic motivation scale (SIMS) | 5 months
  measures younster's motivation to participate the intervention
Toronto Alexitymia Scale (TAS-20) | 5 months
  measures aleksitymia
The Personal Feelings Questionnaire- brief version (PFQ-2 Brief) | 5 months
  measures feelings of quilt

CONTACTS AND LOCATIONS:
Overall Officials: Nina Lindberg, PhD, Principal Investigator — University of Helsinki
Locations (2):
- Finland (2):
  - State Residential Schools, Helsinki
  - Prison and Probation Service of Finland, Helsinki

IPD SHARING:
Plan to Share IPD: No